CLINICAL TRIAL: NCT03421132
Title: The Terry Fox Pan-Canadian Multiple Myeloma Molecular Monitoring Study
Brief Title: Multiple Myeloma Molecular Monitoring Study
Acronym: M4
Status: Active, not recruiting | Type: Observational
Sponsor: Horizon Health Network (Other)
Responsible Party: Principal Investigator, Dr. Anthony Reiman, Principal Investigator, Horizon Health Network
Other Study IDs: M4
Record Dates: First submitted 2018-01-22; First posted 2018-02-05 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human Peripheral Blood: DNA, RNA and WBC.
  Human Bone Marrow: DNA, RNA, WBC, CD138 positive and CD138 negative cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will track 250 multiple myeloma patients across Canada over time, using new lab tests to evaluate their blood and bone marrow, as they receive standard of care treatment. The main hypothesis is that these tests will allow clinicians to better diagnose and manage multiple myeloma, improving patients' quality of life overall.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a deadly cancer of the bone marrow that is challenging to manage and treat: the drugs that are currently available attack the cancer in the same way for everyone, but each patient has different types of MM cancer cells and different family traits that predict better or worse outcomes. As well, the ways in which clinicians test to see if the cancer is in remission are not very good at detecting small numbers of cancer cells still in the bone marrow after treatment - and which will, sooner or later cause the patient to get sick again. The goal of the M4 study is to improve MM patients' survival and quality of life over time, by finding better ways of a) characterizing each patient's experience with the disease, and b) identifying and tracking the small numbers of cells that remain after treatment.

The investigators plan to track 250 patients across Canada over time, who are getting treatment for multiple myeloma. While they are getting treatment, the research team will evaluate samples of their blood and bone marrow with newer, more precise laboratory tests. Participants will also be asked to take part in two scans of their bodies during their treatment. The investigators hypothesize that these tests can help clinicians make better treatment recommendations to patients.

The investigators will look at whether one test is better than another, or if a combination of these tests is needed to have the best information possible to make treatment decisions. At the same time, the research will also explore how and why some patients' cancer becomes resistant to the treatments over time, and how myeloma cells are able to start growing again after treatment. The research team will also collect information on how each patient's health and quality of life changes during and after treatment, and what are the associated costs with these new approaches - to both the healthcare system overall, and to patients.

Once the five-year research program is complete, it is hoped that clinicians will have a new, proven and affordable process of combining these new laboratory tests with the current clinical approach, to create new options to evaluate and treat multiple myeloma.

It is the overall goal that this research will make a difference, right away and across the world, in how doctors treat multiple myeloma, in how it is studied by scientists, and in how patients advocate for their own healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Diagnosed with active multiple myeloma
* Consented to participation in Myeloma Canada Research Network (MCRN) database project
* Previously untreated and eligible for autologous stem-cell transplantation (ASCT)

Exclusion Criteria:

* Ineligible for ASCT
* Does not consent to participate in MCRN database project

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited through hospital oncology clinics across Canada
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Minimal Residual Disease (MRD) Assays | 100 days post-treatment
  Comparison of the sensitivity of two leading-edge MRD assays - (1) multiparameter flow cytometry (MFC), and (2) immunoglobulin gene sequencing (IgS) - in patients who meet the conventional definition of complete remission post-treatment.
Sensitivity of Minimal Residual Disease (MRD) Assays | 12 months post-maintenance therapy
  Comparison of the sensitivity of two leading-edge MRD assays - (1) multiparameter flow cytometry (MFC), and (2) immunoglobulin gene sequencing (IgS) - in patients who meet the conventional definition of complete remission post-treatment.

SECONDARY OUTCOMES:
Comparison of Sensitivity of MRD Assays with PET scans | 12 months post-maintenance therapy
  Comparison of the sensitivity of two MRD assays - (1) multiparameter flow cytometry (MFC), and (2) immunoglobulin gene sequencing (IgS) - with (3) positron emission tomography (PET) imaging scans, in order to determine if PET scans offer additional information above and beyond that offered through the two assays.
Predicting Progression-Free Survival Using MRD Assessment | 5 years
  Establish the prognostic significance of MRD assessment (i.e., the two MRD assays, and PET scans) on progression-free survival
Predicting Overall Survival Using MRD Assessment | 5 years
  Establish the prognostic significance of MRD assessment (i.e., the two MRD assays, and PET scans) on overall survival
Quality-Adjusted Life Years (QALYs) Gained | 5 years
  To fully understand health care costs and benefits associated with personalized risk-adapted testing and monitoring strategies for cancer, compared to current standard of care (e.g., non-personalized), the investigators will create a model that includes cohort's responses on patient-reported health status (using the EuroQol-5D or EQ-5D-L) and use of healthcare resources (using the NCIC Resource Utilization Form), and that will calculate quality-adjusted life years of the participants.
Incremental Cost-Effectiveness of MRD Testing | 5 years
  To fully understand health care costs and benefits associated with personalized risk-adapted testing and monitoring strategies for cancer, compared to current standard of care (e.g., non-personalized), the investigators will create a model that includes cohort's responses on patient-reported health status (using the EuroQol-5D or EQ-5D-L) and use of healthcare resources (using the NCIC Resource Utilization Form), and that will calculate the cost-effectiveness of the MRD assays under investigation.
Productivity Costs Associated with MRD Testing | 5 years
  To fully understand health care costs and benefits associated with personalized risk-adapted testing and monitoring strategies for cancer, compared to current standard of care (e.g., non-personalized), the investigators will create a model that includes cohort's responses on patient-reported health status (using the EuroQol-5D or EQ-5D-L) and use of healthcare resources (using the NCIC Resource Utilization Form), and that will calculate the individual and system-level productivity costs associated with the MRD assays under investigation.
Multiple Myeloma Patients' Quality of Life (QOL) | 5 years
  The investigators will evaluate patients' QOL, especially how it is impacted by treatment, disease and patient characteristics, using a common self-report measure (European Organization for Research and Treatment of Cancer - Quality of Life Questionnaire, or EORTC-QLQ-30). Specific outcomes include QOL at each time point in the study and overall for the cohort, comparing those who achieve MRD and those who do not.
Correlative Study: Sensitivity and Specificity of Drug Resistance Assays | 5 years
  The investigators will also investigate sensitivity and specificity of assays of drug resistance (e.g., why this cancer eventually becomes resistant to the drugs used to treat it)
Correlative Study: Circulating Tumor DNA | 5 years
  The investigators will also investigate prognostic significance of circulating tumour (ct) DNA profiles
Correlative Study: Describing Myeloma Progenitor Populations | 5 years
  The investigators will also seek to understand how the cancer recurs and regrows, even for those who achieve an MRD state.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Reiman, MD, Principal Investigator — Horizon Health Network
Locations (9):
- Canada (9):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital (Horizon Health Network), Saint John, New Brunswick
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Buland Mangukia, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avet-Loiseau H, Corre J, Lauwers-Cances V, Chretien M, Robillard N, Leleu X, et al. 191 Evaluation of Minimal Residual Disease (MRD) By Next Generation Sequencing (NGS) Is Highly Predictive of Progression Free Survival in the IFM/DFCI 2009 Study. Blood 126(23): 191, 2015.
- [Background] Benboubker L, Dimopoulos MA, Dispenzieri A, Catalano J, Belch AR, Cavo M, Pinto A, Weisel K, Ludwig H, Bahlis N, Banos A, Tiab M, Delforge M, Cavenagh J, Geraldes C, Lee JJ, Chen C, Oriol A, de la Rubia J, Qiu L, White DJ, Binder D, Anderson K, Fermand JP, Moreau P, Attal M, Knight R, Chen G, Van Oostendorp J, Jacques C, Ervin-Haynes A, Avet-Loiseau H, Hulin C, Facon T; FIRST Trial Team. Lenalidomide and dexamethasone in transplant-ineligible patients with myeloma. N Engl J Med. 2014 Sep 4;371(10):906-17. doi: 10.1056/NEJMoa1402551. PMID 25184863
- [Background] Bolli N, Avet-Loiseau H, Wedge DC, Van Loo P, Alexandrov LB, Martincorena I, Dawson KJ, Iorio F, Nik-Zainal S, Bignell GR, Hinton JW, Li Y, Tubio JM, McLaren S, O' Meara S, Butler AP, Teague JW, Mudie L, Anderson E, Rashid N, Tai YT, Shammas MA, Sperling AS, Fulciniti M, Richardson PG, Parmigiani G, Magrangeas F, Minvielle S, Moreau P, Attal M, Facon T, Futreal PA, Anderson KC, Campbell PJ, Munshi NC. Heterogeneity of genomic evolution and mutational profiles in multiple myeloma. Nat Commun. 2014;5:2997. doi: 10.1038/ncomms3997. PMID 24429703
- [Background] Chapman MA, Lawrence MS, Keats JJ, Cibulskis K, Sougnez C, Schinzel AC, Harview CL, Brunet JP, Ahmann GJ, Adli M, Anderson KC, Ardlie KG, Auclair D, Baker A, Bergsagel PL, Bernstein BE, Drier Y, Fonseca R, Gabriel SB, Hofmeister CC, Jagannath S, Jakubowiak AJ, Krishnan A, Levy J, Liefeld T, Lonial S, Mahan S, Mfuko B, Monti S, Perkins LM, Onofrio R, Pugh TJ, Rajkumar SV, Ramos AH, Siegel DS, Sivachenko A, Stewart AK, Trudel S, Vij R, Voet D, Winckler W, Zimmerman T, Carpten J, Trent J, Hahn WC, Garraway LA, Meyerson M, Lander ES, Getz G, Golub TR. Initial genome sequencing and analysis of multiple myeloma. Nature. 2011 Mar 24;471(7339):467-72. doi: 10.1038/nature09837. PMID 21430775
- [Background] Chng WJ, Dispenzieri A, Chim CS, Fonseca R, Goldschmidt H, Lentzsch S, Munshi N, Palumbo A, Miguel JS, Sonneveld P, Cavo M, Usmani S, Durie BG, Avet-Loiseau H; International Myeloma Working Group. IMWG consensus on risk stratification in multiple myeloma. Leukemia. 2014 Feb;28(2):269-77. doi: 10.1038/leu.2013.247. Epub 2013 Aug 26. PMID 23974982
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Gonzalez D, van der Burg M, Garcia-Sanz R, Fenton JA, Langerak AW, Gonzalez M, van Dongen JJ, San Miguel JF, Morgan GJ. Immunoglobulin gene rearrangements and the pathogenesis of multiple myeloma. Blood. 2007 Nov 1;110(9):3112-21. doi: 10.1182/blood-2007-02-069625. Epub 2007 Jul 18. PMID 17634408
- [Background] Kapoor P, Kumar SK, Dispenzieri A, Lacy MQ, Buadi F, Dingli D, Russell SJ, Hayman SR, Witzig TE, Lust JA, Leung N, Lin Y, Zeldenrust SR, McCurdy A, Greipp PR, Kyle RA, Rajkumar SV, Gertz MA. Importance of achieving stringent complete response after autologous stem-cell transplantation in multiple myeloma. J Clin Oncol. 2013 Dec 20;31(36):4529-35. doi: 10.1200/JCO.2013.49.0086. Epub 2013 Nov 18. PMID 24248686
- [Background] Korde N, Roschewski M, Zingone A, Kwok M, Manasanch EE, Bhutani M, Tageja N, Kazandjian D, Mailankody S, Wu P, Morrison C, Costello R, Zhang Y, Burton D, Mulquin M, Zuchlinski D, Lamping L, Carpenter A, Wall Y, Carter G, Cunningham SC, Gounden V, Sissung TM, Peer C, Maric I, Calvo KR, Braylan R, Yuan C, Stetler-Stevenson M, Arthur DC, Kong KA, Weng L, Faham M, Lindenberg L, Kurdziel K, Choyke P, Steinberg SM, Figg W, Landgren O. Treatment With Carfilzomib-Lenalidomide-Dexamethasone With Lenalidomide Extension in Patients With Smoldering or Newly Diagnosed Multiple Myeloma. JAMA Oncol. 2015 Sep;1(6):746-54. doi: 10.1001/jamaoncol.2015.2010. PMID 26181891
- [Background] Kumar S, Paiva B, Anderson KC, Durie B, Landgren O, Moreau P, Munshi N, Lonial S, Blade J, Mateos MV, Dimopoulos M, Kastritis E, Boccadoro M, Orlowski R, Goldschmidt H, Spencer A, Hou J, Chng WJ, Usmani SZ, Zamagni E, Shimizu K, Jagannath S, Johnsen HE, Terpos E, Reiman A, Kyle RA, Sonneveld P, Richardson PG, McCarthy P, Ludwig H, Chen W, Cavo M, Harousseau JL, Lentzsch S, Hillengass J, Palumbo A, Orfao A, Rajkumar SV, Miguel JS, Avet-Loiseau H. International Myeloma Working Group consensus criteria for response and minimal residual disease assessment in multiple myeloma. Lancet Oncol. 2016 Aug;17(8):e328-e346. doi: 10.1016/S1470-2045(16)30206-6. PMID 27511158
- [Background] Leung-Hagesteijn C, Erdmann N, Cheung G, Keats JJ, Stewart AK, Reece DE, Chung KC, Tiedemann RE. Xbp1s-Negative Tumor B Cells and Pre-Plasmablasts Mediate Therapeutic Proteasome Inhibitor Resistance in Multiple Myeloma. Cancer Cell. 2015 Oct 12;28(4):541-542. doi: 10.1016/j.ccell.2015.09.010. Epub 2015 Oct 12. No abstract available. PMID 28854350
- [Background] Mailankody S, Korde N, Lesokhin AM, Lendvai N, Hassoun H, Stetler-Stevenson M, Landgren O. Minimal residual disease in multiple myeloma: bringing the bench to the bedside. Nat Rev Clin Oncol. 2015 May;12(5):286-95. doi: 10.1038/nrclinonc.2014.239. Epub 2015 Jan 27. PMID 25622976
- [Background] Martinez-Lopez J, Lahuerta JJ, Pepin F, Gonzalez M, Barrio S, Ayala R, Puig N, Montalban MA, Paiva B, Weng L, Jimenez C, Sopena M, Moorhead M, Cedena T, Rapado I, Mateos MV, Rosinol L, Oriol A, Blanchard MJ, Martinez R, Blade J, San Miguel J, Faham M, Garcia-Sanz R. Prognostic value of deep sequencing method for minimal residual disease detection in multiple myeloma. Blood. 2014 May 15;123(20):3073-9. doi: 10.1182/blood-2014-01-550020. Epub 2014 Mar 19. PMID 24646471
- [Background] Matsui W, Wang Q, Barber JP, Brennan S, Smith BD, Borrello I, McNiece I, Lin L, Ambinder RF, Peacock C, Watkins DN, Huff CA, Jones RJ. Clonogenic multiple myeloma progenitors, stem cell properties, and drug resistance. Cancer Res. 2008 Jan 1;68(1):190-7. doi: 10.1158/0008-5472.CAN-07-3096. PMID 18172311
- [Background] Moreau P, Attal M, Caillot D, Macro M, Karlin L, Garderet L, Facon T, Benboubker L, Escoffre-Barbe M, Stoppa AM, Laribi K, Hulin C, Perrot A, Marit G, Eveillard JR, Caillon F, Bodet-Milin C, Pegourie B, Dorvaux V, Chaleteix C, Anderson K, Richardson P, Munshi NC, Avet-Loiseau H, Gaultier A, Nguyen JM, Dupas B, Frampas E, Kraeber-Bodere F. Prospective Evaluation of Magnetic Resonance Imaging and [18F]Fluorodeoxyglucose Positron Emission Tomography-Computed Tomography at Diagnosis and Before Maintenance Therapy in Symptomatic Patients With Multiple Myeloma Included in the IFM/DFCI 2009 Trial: Results of the IMAJEM Study. J Clin Oncol. 2017 Sep 1;35(25):2911-2918. doi: 10.1200/JCO.2017.72.2975. Epub 2017 Jul 7. PMID 28686535
- [Background] Nygaard AD, Garm Spindler KL, Pallisgaard N, Andersen RF, Jakobsen A. The prognostic value of KRAS mutated plasma DNA in advanced non-small cell lung cancer. Lung Cancer. 2013 Mar;79(3):312-7. doi: 10.1016/j.lungcan.2012.11.016. Epub 2012 Dec 11. PMID 23238036
- [Background] Paiva B, Vidriales MB, Cervero J, Mateo G, Perez JJ, Montalban MA, Sureda A, Montejano L, Gutierrez NC, Garcia de Coca A, de Las Heras N, Mateos MV, Lopez-Berges MC, Garcia-Boyero R, Galende J, Hernandez J, Palomera L, Carrera D, Martinez R, de la Rubia J, Martin A, Blade J, Lahuerta JJ, Orfao A, San Miguel JF; GEM (Grupo Espanol de MM)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Groups. Multiparameter flow cytometric remission is the most relevant prognostic factor for multiple myeloma patients who undergo autologous stem cell transplantation. Blood. 2008 Nov 15;112(10):4017-23. doi: 10.1182/blood-2008-05-159624. Epub 2008 Jul 31. PMID 18669875
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Rawstron AC, Child JA, de Tute RM, Davies FE, Gregory WM, Bell SE, Szubert AJ, Navarro-Coy N, Drayson MT, Feyler S, Ross FM, Cook G, Jackson GH, Morgan GJ, Owen RG. Minimal residual disease assessed by multiparameter flow cytometry in multiple myeloma: impact on outcome in the Medical Research Council Myeloma IX Study. J Clin Oncol. 2013 Jul 10;31(20):2540-7. doi: 10.1200/JCO.2012.46.2119. Epub 2013 Jun 3. PMID 23733781
- [Background] Rawstron AC, Gregory WM, de Tute RM, Davies FE, Bell SE, Drayson MT, Cook G, Jackson GH, Morgan GJ, Child JA, Owen RG. Minimal residual disease in myeloma by flow cytometry: independent prediction of survival benefit per log reduction. Blood. 2015 Mar 19;125(12):1932-5. doi: 10.1182/blood-2014-07-590166. Epub 2015 Feb 2. PMID 25645353
- [Background] Reinert T, Scholer LV, Thomsen R, Tobiasen H, Vang S, Nordentoft I, Lamy P, Kannerup AS, Mortensen FV, Stribolt K, Hamilton-Dutoit S, Nielsen HJ, Laurberg S, Pallisgaard N, Pedersen JS, Orntoft TF, Andersen CL. Analysis of circulating tumour DNA to monitor disease burden following colorectal cancer surgery. Gut. 2016 Apr;65(4):625-34. doi: 10.1136/gutjnl-2014-308859. Epub 2015 Feb 4. PMID 25654990
- [Background] Roschewski M, Dunleavy K, Pittaluga S, Moorhead M, Pepin F, Kong K, Shovlin M, Jaffe ES, Staudt LM, Lai C, Steinberg SM, Chen CC, Zheng J, Willis TD, Faham M, Wilson WH. Circulating tumour DNA and CT monitoring in patients with untreated diffuse large B-cell lymphoma: a correlative biomarker study. Lancet Oncol. 2015 May;16(5):541-9. doi: 10.1016/S1470-2045(15)70106-3. Epub 2015 Apr 1. PMID 25842160
- [Background] Schwarzenbach H, Eichelser C, Kropidlowski J, Janni W, Rack B, Pantel K. Loss of heterozygosity at tumor suppressor genes detectable on fractionated circulating cell-free tumor DNA as indicator of breast cancer progression. Clin Cancer Res. 2012 Oct 15;18(20):5719-30. doi: 10.1158/1078-0432.CCR-12-0142. Epub 2012 Sep 25. PMID 23014523
- [Background] Schwarzenbach H, Hoon DS, Pantel K. Cell-free nucleic acids as biomarkers in cancer patients. Nat Rev Cancer. 2011 Jun;11(6):426-37. doi: 10.1038/nrc3066. Epub 2011 May 12. PMID 21562580
- [Background] Silva JM, Silva J, Sanchez A, Garcia JM, Dominguez G, Provencio M, Sanfrutos L, Jareno E, Colas A, Espana P, Bonilla F. Tumor DNA in plasma at diagnosis of breast cancer patients is a valuable predictor of disease-free survival. Clin Cancer Res. 2002 Dec;8(12):3761-6. PMID 12473587
- [Background] Vij R, Mazumder A, Klinger M, O'Dea D, Paasch J, Martin T, Weng L, Park J, Fiala M, Faham M, Wolf J. Deep sequencing reveals myeloma cells in peripheral blood in majority of multiple myeloma patients. Clin Lymphoma Myeloma Leuk. 2014 Apr;14(2):131-139.e1. doi: 10.1016/j.clml.2013.09.013. Epub 2013 Oct 2. PMID 24629890
- [Background] Zamagni E, Nanni C, Mancuso K, Tacchetti P, Pezzi A, Pantani L, Zannetti B, Rambaldi I, Brioli A, Rocchi S, Terragna C, Martello M, Marzocchi G, Borsi E, Rizzello I, Fanti S, Cavo M. PET/CT Improves the Definition of Complete Response and Allows to Detect Otherwise Unidentifiable Skeletal Progression in Multiple Myeloma. Clin Cancer Res. 2015 Oct 1;21(19):4384-90. doi: 10.1158/1078-0432.CCR-15-0396. Epub 2015 Jun 15. PMID 26078390

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT03421132/Prot_SAP_000.pdf